CLINICAL TRIAL: NCT00924066
Title: A Phase II Clinical Trial of Ixabepilone (Ixempra [R], BMS-247550, NSC 710428), an Epothilone B Analog, in Cervical Cancer
Brief Title: Ixabepilone to Treat Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature closure due to slow/insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Antonio Fojo, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090037; 09-C-0037; NCT00798928 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Cervical Carcinoma; Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Carcinoma, Non-SquamousType
Keywords: Ixabepilone; BMS-247550; Ixempra; Cervical Cancer; Epothilone
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Squamous and Nonsquamous participants (Experimental): Squamous cell carcinoma is a histologic subtype of cervical cancer. Squamous cell carcinoma of the cervix (80%) is much more common than adenocarcinoma of the cervix.
  Non squamous carcinoma is a histologic subtype of cervical cancer. It is the second most common form of cervical cancer; consists of adenocarcinoma, adenosquamous and non squamous (not otherwise specified) subtypes.
  All participants in both arms received ixabepilone 6 mg/m^2 x 5 days, each cycle.
  Interventions: Drug: Ixempra (Ixabepilone (BMS-247550) )

INTERVENTIONS:
Drug: Ixempra (Ixabepilone (BMS-247550) ) — Participants received Ixabepilone 6mg/m^2 for a total of 30mg/m^2 inpatient or outpatient intravenously over an hour on the first five days of each 21 day cycle.
  Other Names: BMS-247550

SUMMARY:
Background:

* Ixabepilone is a member of the class of drugs called epothilones. These drugs interfere with the ability of cancer cells to replicate.
* Epothilones are similar to taxanes, another class of drugs, which includes the drug Taxol. Taxol is widely used to treat a variety of cancers.
* Ixabepilone can work in cells that are resistant to Taxol.

Objectives:

* To determine whether ixabepilone is effective for treating cervical cancer.

Eligibility:

* Women 18 years of age or older with cervical cancer.

Design:

* Patients receive ixabepilone intravenously (through a vein) over 60 minutes on the first 5 days of each 21-day treatment cycle. Their dosage may be adjusted according to how their bodies respond to the drug.
* The number of cycles each woman receives depends on her response to the treatment.
* Patients have CT (computed tomography) scans and other tests before starting treatment and then every other treatment cycle to determine the response of the tumor to ixabepilone.
* Patients who can undergo a tumor biopsy (surgical removal of a sample of tumor tissue) are asked to have a biopsy done before starting treatment with ixabepilone and again on the fourth or fifth day of treatment. This procedure is optional.

DETAILED DESCRIPTION:
Background

* Ixabepilone (Ixempra (Trademark), BMS-247550, NSC 710428) is a semi-synthetic analog of the natural product epothilone B.
* The epothilones are a novel class of non-taxane microtubule-stabilizing agents obtained from the fermentation of the cellulose degrading myxobacteria, Sorangium cellulosum.
* Ixabepilone is active against cancer models that are naturally insensitive to paclitaxel or have developed resistance to paclitaxel, both in-vitro and in-vivo.

Objectives

Primary-

- Establish the efficacy of the investigational agent ixabepilone in patients with cervical carcinoma when administered as a daily one-hour infusion on days 1 to 5 every three weeks, as measured by overall response (PR (partial response) +CR (complete response)).

Secondary-

* Assess pharmacodynamic endpoints to determine the extent of tubulin polymerization and whether or not there has been activation of cellular death pathways distal to the target.
* Estimate progression-free survival and duration of response.

Eligibility

* Age greater than 18
* Histologic or cytologic confirmation of cervical carcinoma; either squamous cell or non-squamous consisting of cervical adenocarcinoma, cervical adenosquamous carcinoma or cervical carcinoma, non-squamous type.

Design

* Phase II study, open, non-randomized
* Ixabepilone will be administered at a dose of 6mg/m^2 daily on days 1 through 5, every three weeks.
* Restaging will be done every two cycles using RECIST (Response Evaluation Criteria in Solid Tumors)
* Planned maximum enrollment 76 persons

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must fulfill all of the following criteria to be eligible for study admission:

1. Age greater than or equal to 18 years.
2. Histologic or cytologic confirmation of cervical carcinoma, squamous or non-squamous. Within the non-squamous cohort is adenocarcinoma and adenosquamous as well as non-squamous (not otherwise specified).
3. Subjects with unresectable recurrent cervical cancer are eligible.
4. Measurable disease that can be assessed using RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
5. Performance Status ECOG (Eastern Cooperative Oncology Group) 0-2.
6. Life expectancy of 3 months or greater.
7. Suitable candidate for receiving planned therapy as evidenced by screening laboratory assessments of hematologic, renal, hepatic, and metabolic functions: platelet count greater than or equal to 75,000/mm^3, absolute granulocyte count (AGC) greater than or equal to 1,000/mm^3, serum creatinine less than or equal to 1.6 or a measured creatinine clearance greater than or equal to 40 ml/min, SGPT (serum glutamic pyruvic transaminase) and SGOT (serum glutamic oxaloacetic transaminase) less than or equal to 2.5 times the NL (normal limit), and total bilirubin less than or equal to 1.5 times the NL (in patients with clinical evidence of Gilberts' disease, less than or equal to 3 times the NL).

   Note: A diagnosis of Gilbert s disease will be made in the presence of (1) unconjugated hyperbilirubinemia noted on several occasions; (2) normal results from CBC (complete blood count) count, reticulocyte count, and blood smear; (3) normal liver function test results; and (4) an absence of other disease processes that can explain the unconjugated hyperbilirubinemia.
8. Greater than or equal to 4 weeks from prior radiation, intravenous chemotherapy or immunotherapy; greater than or equal to 6 weeks from prior nitrosourea; greater than or equal to 2 weeks from a prior phase 0 study .
9. No serious intercurrent medical illness.
10. The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol.
11. Prior therapy with cisplatin or carboplatin is required.

EXCLUSION CRITERIA:

Patients with any of the following will be excluded from study entry:

1. Pregnant or nursing women are not eligible; neither are women of childbearing potential unless using effective contraception as determined by the patients physician.
2. Patients with a history of CNS (central nervous system) metastases, because symptoms/signs of progressive disease may be confused with drug-related toxicities, unless control has been achieved with either radiation or surgical resection at least three months prior to enrollment on study.
3. Patients who are poor medical risk because of other non malignant systemic disease or active, uncontrolled infection.
4. Human Immunodeficiency Virus (HIV) positive patients will be considered for eligibility, as long as they are not receiving antiretroviral drugs with strong CYP3A4 (cytochrome P450 3A4) inhibitory activity.
5. Prior craniospinal radiation, or total body irradiation (TBI).
6. Patients receiving other investigational drugs, or strong CYP3A3 inhibitors (see Section 3.6 for details) that cannot be discontinued or substituted.
7. CTCAE (Common Terminology Criteria for Adverse Events) Grade 2 or greater motor or sensory neuropathy.
8. Known prior severe hypersensitivity reactions to agents containing Cremophor (Trademark) EL.
9. Women with localized disease who are potentially curable through surgical resection.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio T Fojo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkin DM, Laara E, Muir CS. Estimates of the worldwide frequency of sixteen major cancers in 1980. Int J Cancer. 1988 Feb 15;41(2):184-97. doi: 10.1002/ijc.2910410205. PMID 3338870
- [Background] Leveque J, Laurent JF, Burtin F, Foucher F, Goyat F, Grall JY, Meunier B. Prognostic factors of the uterine cervix adenocarcinoma. Eur J Obstet Gynecol Reprod Biol. 1998 Oct;80(2):209-14. doi: 10.1016/s0301-2115(98)00106-7. PMID 9846671
- [Background] Alfsen GC, Kristensen GB, Skovlund E, Pettersen EO, Abeler VM. Histologic subtype has minor importance for overall survival in patients with adenocarcinoma of the uterine cervix: a population-based study of prognostic factors in 505 patients with nonsquamous cell carcinomas of the cervix. Cancer. 2001 Nov 1;92(9):2471-83. doi: 10.1002/1097-0142(20011101)92:93.0.co;2-k. PMID 11745305
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0037.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Squamous and Nonsquamous Participants
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Squamous and Nonsquamous Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.79 (9.17)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Tumor Response (PR + CR) Per RECIST
Description: Establish the efficacy of the investigational agent Ixabepilone in patients with cervical carcinoma per the Response Evaluation Criteria in Solid Tumors (RECIST) when Ixabepilone is administered as a daily 1 hour infusion on days 1-5 every 3 weeks. Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Not evaluable (NE) means the participant was not evaluable because there was not a scan available to compare to the baseline scan.
Time Frame: Every 6 weeks, up to 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Squamous and Nonsquamous Participants
Number analyzed (Participants) | 41
Participants
  Not Evaluable (only 1 cycle) | 2
  Progressive Disease | 25
  Stable Disease | 10
  Partial Response | 4
  Complete Response | 0

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 61 months
Population: Adverse events are grouped together because the histology cohort has no bearing on the adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Squamous and Nonsquamous Participants
Number analyzed (Participants) | 41
Participants | 41

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 61 months.
Groups:
- Adverse Events for Squamous and Non-squamous Participants: Squamous cell carcinoma is a histologic subtype of cervical cancer. Squamous cell carcinoma of the cervix (80%) is much more common than adenocarcinoma of the cervix.
  Non squamous carcinoma is a histologic subtype of cervical cancer. It is the second most common form of cervical cancer; consists of adenocarcinoma, adenosquamous and non squamous (not otherwise specified) subtypes.
  All participants in both arms received ixabepilone 6 mg/m^2 x 5 days, each cycle.
Arm/Group | Adverse Events for Squamous and Non-squamous Participants
All-Cause Mortality (participants affected / at risk) | 2/41
Serious Adverse Events (participants affected / at risk) | 18/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events for Squamous and Non-squamous Participants (N=41)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Enterocolitis infectious (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileal fistula (Gastrointestinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized pain
Nausea (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Phlebitis infective (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Urinary fistula (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events for Squamous and Non-squamous Participants (N=41)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (26)
Alkaline phosphatase increased (Investigations) | 21 (44)
Allergic reaction (Immune system disorders) | 3 (3)
Allergic rhinitis (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (14)
Anemia (Blood and lymphatic system disorders) | 41 (256)
Anorexia (Metabolism and nutrition disorders) | 19 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11)
Aspartate aminotransferase increased (Investigations) | 14 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Blood bilirubin increased (Investigations) | 5 (10)
Blurred vision (Eye disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
CPK increased (Investigations) | 4 (5)
Chills (General disorders) | 3 (3)
Colonic fistula (Gastrointestinal disorders) | 1 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 12 (31)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 13 (21)
Dizziness (Nervous system disorders) | 6 (6)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Edema limbs (General disorders) | 9 (12)
Edema trunk (General disorders) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 23 (46)
Fever (General disorders) | 8 (14)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Hematuria (Renal and urinary disorders) | 5 (5)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 15 (35)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (9)
Hypernatremia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Vascular disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 12 (24)
Hypoalbuminemia (Metabolism and nutrition disorders) | 31 (92)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (18)
Hypokalemia (Metabolism and nutrition disorders) | 18 (41)
Hypomagnesemia (Metabolism and nutrition disorders) | 25 (79)
Hyponatremia (Metabolism and nutrition disorders) | 22 (48)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (32)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Infections and infestations - Other, specify (Toe nail W normal ANC) (Infections and infestations) | 2 (2)
Infusion related reaction (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (3)
Investigations - Other, specify (Investigations) | 4 (6)
Lymphocyte count decreased (Investigations) | 41 (304)
Mucosal infection (Infections and infestations) | 3 (3)
Mucositis oral (General disorders) | 6 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 25 (46)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 4 (5)
Neutrophil count decreased (Investigations) | 8 (12)
Non-cardiac chest pain (General disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Pelvic pain (Reproductive system and breast disorders) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (14)
Platelet count decreased (Investigations) | 25 (83)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal mucositis (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — Surgery to create a colostomy
Syncope (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Urinary fistula (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (8)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 3 (5)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (32)
Weight loss (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 18 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-02-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT00924066/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT00924066/ICF_001.pdf